CLINICAL TRIAL: NCT06958666
Title: Effectiveness of DITM Versus IMT in COPD Patients With High Symptom Burden and High Risk of Acute Exacerbation: A Randomized Controlled Study
Brief Title: Effectiveness of DITM Versus IMT in COPD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Collaborators: Jingyao (Hangzhou) Health Technology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Huiqing Ge, Director of Respiratory Therapy Department, Sir Run Run Shaw Hospital, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20250119
Record Dates: First submitted 2025-04-16; First posted 2025-05-06 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: Pulmonary Rehabilitation; COPD; GOLD2024; Global Initiative for Chronic Obstructive Lung Disease; Digital Inhaled Therapy Management; Inspiratory Muscle Training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Digital Inhalation Management Group (Experimental): Digital Inhalation Management Group will receive digital inhaled therapy management only
  Interventions: Device: Digital Inhaled Therapy Management
- Inspiratory Muscle Training Group (Experimental): Inspiratory Muscle Training Group will receive inspiratory muscle training only
  Interventions: Device: Inspiratory Muscle Training
- Inhalation Muscle Training Combined with Digital Inhalation Therapy Management Group (Experimental): The subjects will receive Inspiratory muscle training equipment, ancillary software, inspiratory muscle training plan, and equipment user guide in addition to training on the use of Digital Inhalation Administration device.
  Interventions: Device: Digital Inhaled Therapy Management; Device: Inspiratory Muscle Training
- Compare Group (No Intervention): The subjects will receive standardized verbal training and demonstration of inhalation techniques. No additional equipment provided

INTERVENTIONS:
Device: Digital Inhaled Therapy Management — The subjects will be trained on their inhalation techniques with the "Digital Medication Administration Device" consists of an inhalation device with a display and inhalation technique assessment module. The device will show a standardized video demonstration and will evaluate the subjects' inhalation technique. A printed report will be available afterwards.
  A home-based inhalation management service package will be provided to the subjects including a digital sensor that records the time, frequency, and key inhalation technique parameters for each use of metered-dose inhalers or dry powder inhalers, and automatically synchronizes the data to the cloud. The data is then analyzed for adherence and technique performance. Based on the data, subjects will receive medication reminders and voice alerts for any technique errors on the app provided with the package. Visual charts of medication adherence and inhalation technique will be available to reinforce self-management.
  Arms: Digital Inhalation Management Group; Inhalation Muscle Training Combined with Digital Inhalation Therapy Management Group
Device: Inspiratory Muscle Training — The subjects will receive standardized verbal training and demonstration of inhalation techniques and any questions will be answered Inspiratory muscle training equipment, ancillary software, inspiratory muscle training plan, and equipment user guide will be sent home with the patient.
  Arms: Inhalation Muscle Training Combined with Digital Inhalation Therapy Management Group; Inspiratory Muscle Training Group

SUMMARY:
The goal of this clinical trial is to learn if digital inhaled therapy management (DITM) and inspiratory muscle training (IMT), alone or in combination, can improve outcomes in adults aged 40 years and older with symptomatic, high-risk chronic obstructive pulmonary disease (COPD) with moderate to severe airflow limitation (FEV1/FVC < 60%). The main questions it aims to answer are:

Does DITM reduce the rate of moderate to severe COPD exacerbations and hospitalizations compared to usual care? Does IMT reduce the rate of moderate to severe COPD exacerbations and hospitalizations compared to usual care? Does the combination of DITM and IMT reduce the rate of moderate to severe COPD exacerbations and hospitalizations compared to usual care? What are the effects of DITM, IMT, and their combination on the time to first moderate to severe exacerbation, COPD Assessment Test (CAT) score, modified Medical Research Council (mMRC) score, and St. George's Respiratory Questionnaire for chronic obstructive pulmonary disease (SGRQ-C) score? Researchers will compare four groups: a DITM group, an IMT group, a DITM+IMT group, and a control group receiving usual care, to see if these interventions improve outcomes related to COPD exacerbations, symptoms, quality of life, and inspiratory muscle strength.

Participants will:

DITM Group: Receive training on inhaler technique using a digital device and use a digital sensor with a mobile app for home-based inhalation management, including reminders and feedback.

IMT Group: Receive verbal inhaler technique training and use a breathing trainer with accompanying software for inspiratory muscle training.

DITM+IMT Group: Receive both the digital inhalation management and inspiratory muscle training interventions.

Control Group: Receive verbal inhaler technique training only. All participants will undergo baseline assessments and follow-up assessments at 3, 6, and 12 months, including questionnaires, lung function tests, respiratory muscle strength measurements, and a 6-minute walk test. They will also report on any COPD exacerbations experienced during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as COPD according to "GOLD2024"
* Lung function results FEV1/FVC<60%
* Patients with stable COPD who meet one of the following criteria: (A)with CAT score ≥10 or mMRC≥2; (B) ≥2 moderate acute exacerbation or ≥1 hospitalization in the past 12 months
* Uses Budesonide MDI (Breztri Aerosphere) or Fluticasone, umeclidinium, and vilanterol (Trelegy Ellipta) or umeclidinium and vilanterol (Anoro Ellipta) as maintenance drug for COPD management
* Volunteer to participate in this study and sign the informed consent form. If the subject is unable to read and sign the informed consent form due to incapacity, his/her guardian shall act on his/her behalf to read and sign the informed consent form.

Exclusion Criteria:

* Unstable angina or severe arrhythmia
* Severe weakness-related fatigue, such as in advanced congestive heart failure or chemotherapy-related fatigue
* Unstable mental illness with a risk of self-harm or harm to others
* Severe cognitive impairment, progressive neuromuscular disease
* Pregnant and breastfeeding women
* Life expectancy of less than 6 months
* Pregnant and breastfeeding women
* Inability to cooperate with pulmonary function tests
* Inability to complete the entire follow-up period
* Vulnerable populations other than the elderly, including individuals with mental illness, cognitive impairment, critically ill patients, illiterate individuals, etc.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Rate of acute exacerbation of moderate-to-severe COPD and hospitalization during follow-up period | Follow-up assessments are collected 3 months, 6 months, and 12 months after their initial training
  Rate of acute exacerbation of moderate-to-severe COPD and hospitalization during follow-up period will be accessed as the primary endpoint. Acute exacerbation of COPD is defined according to the "Chinese Expert Consensus on the Diagnosis and Treatment of Acute Exacerbation of COPD" 2023 version.

SECONDARY OUTCOMES:
Days to first Moderate-to-Severe Acute Exacerbation | Follow-up assessments are collected 3 months, 6 months, and 12 months after their initial training
  Time from baseline to the occurrence of the first acute exacerbation in days.
COPD Assessment Test (CAT) Score | Follow-up assessments are collected 3 months, 6 months, and 12 months after their initial training
  Self-reported measure of health status in COPD patients, assessed using the CAT questionnaire. Higher scores indicate a greater impact of COPD on daily life.
Modified Medical Research Council (mMRC) Dyspnea Score | Follow-up assessments are collected 3 months, 6 months, and 12 months after their initial training
  Patient-rated scale assessing the severity of breathlessness. Higher grade indicates higher severity.
St. George's Respiratory Questionnaire (SGRQ) Score | assessed only during the last two follow ups (6 months and 12 months).
  Quality of life assessment specific to respiratory diseases. Higher scores reflect worse health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Huiqing Ge, MD, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Molimard M, Raherison C, Lignot S, Balestra A, Lamarque S, Chartier A, Droz-Perroteau C, Lassalle R, Moore N, Girodet PO. Chronic obstructive pulmonary disease exacerbation and inhaler device handling: real-life assessment of 2935 patients. Eur Respir J. 2017 Feb 15;49(2):1601794. doi: 10.1183/13993003.01794-2016. Print 2017 Feb. PMID 28182569
- [Background] Melani AS, Bonavia M, Cilenti V, Cinti C, Lodi M, Martucci P, Serra M, Scichilone N, Sestini P, Aliani M, Neri M; Gruppo Educazionale Associazione Italiana Pneumologi Ospedalieri. Inhaler mishandling remains common in real life and is associated with reduced disease control. Respir Med. 2011 Jun;105(6):930-8. doi: 10.1016/j.rmed.2011.01.005. Epub 2011 Mar 2. PMID 21367593
- [Background] Molimard M, Raherison C, Lignot S, Depont F, Abouelfath A, Moore N. Assessment of handling of inhaler devices in real life: an observational study in 3811 patients in primary care. J Aerosol Med. 2003 Fall;16(3):249-54. doi: 10.1089/089426803769017613. PMID 14572322
- [Background] Cho-Reyes S, Celli BR, Dembek C, Yeh K, Navaie M. Inhalation Technique Errors with Metered-Dose Inhalers Among Patients with Obstructive Lung Diseases: A Systematic Review and Meta-Analysis of U.S. Studies. Chronic Obstr Pulm Dis. 2019 Jul 24;6(3):267-280. doi: 10.15326/jcopdf.6.3.2018.0168. PMID 31342732
- [Background] Sanchis J, Gich I, Pedersen S; Aerosol Drug Management Improvement Team (ADMIT). Systematic Review of Errors in Inhaler Use: Has Patient Technique Improved Over Time? Chest. 2016 Aug;150(2):394-406. doi: 10.1016/j.chest.2016.03.041. Epub 2016 Apr 7. PMID 27060726
- [Background] Crompton GK, Barnes PJ, Broeders M, Corrigan C, Corbetta L, Dekhuijzen R, Dubus JC, Magnan A, Massone F, Sanchis J, Viejo JL, Voshaar T; Aerosol Drug Management Improvement Team. The need to improve inhalation technique in Europe: a report from the Aerosol Drug Management Improvement Team. Respir Med. 2006 Sep;100(9):1479-94. doi: 10.1016/j.rmed.2006.01.008. Epub 2006 Feb 21. PMID 16495040
- [Background] Souza ML, Meneghini AC, Ferraz E, Vianna EO, Borges MC. Knowledge of and technique for using inhalation devices among asthma patients and COPD patients. J Bras Pneumol. 2009 Sep;35(9):824-31. doi: 10.1590/s1806-37132009000900002. English, Portuguese. PMID 19820807
- [Background] Raissy HH, Kelly HW, Harkins M, Szefler SJ. Inhaled corticosteroids in lung diseases. Am J Respir Crit Care Med. 2013 Apr 15;187(8):798-803. doi: 10.1164/rccm.201210-1853PP. PMID 23370915
- [Background] Chen S, Kuhn M, Prettner K, Yu F, Yang T, Barnighausen T, Bloom DE, Wang C. The global economic burden of chronic obstructive pulmonary disease for 204 countries and territories in 2020-50: a health-augmented macroeconomic modelling study. Lancet Glob Health. 2023 Aug;11(8):e1183-e1193. doi: 10.1016/S2214-109X(23)00217-6. PMID 37474226
- [Background] Meghji J, Mortimer K, Agusti A, Allwood BW, Asher I, Bateman ED, Bissell K, Bolton CE, Bush A, Celli B, Chiang CY, Cruz AA, Dinh-Xuan AT, El Sony A, Fong KM, Fujiwara PI, Gaga M, Garcia-Marcos L, Halpin DMG, Hurst JR, Jayasooriya S, Kumar A, Lopez-Varela MV, Masekela R, Mbatchou Ngahane BH, Montes de Oca M, Pearce N, Reddel HK, Salvi S, Singh SJ, Varghese C, Vogelmeier CF, Walker P, Zar HJ, Marks GB. Improving lung health in low-income and middle-income countries: from challenges to solutions. Lancet. 2021 Mar 6;397(10277):928-940. doi: 10.1016/S0140-6736(21)00458-X. Epub 2021 Feb 22. PMID 33631128
- [Background] Zhou M, Wang H, Zeng X, Yin P, Zhu J, Chen W, Li X, Wang L, Wang L, Liu Y, Liu J, Zhang M, Qi J, Yu S, Afshin A, Gakidou E, Glenn S, Krish VS, Miller-Petrie MK, Mountjoy-Venning WC, Mullany EC, Redford SB, Liu H, Naghavi M, Hay SI, Wang L, Murray CJL, Liang X. Mortality, morbidity, and risk factors in China and its provinces, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 Sep 28;394(10204):1145-1158. doi: 10.1016/S0140-6736(19)30427-1. Epub 2019 Jun 24. PMID 31248666
- [Background] Wang C, Xu J, Yang L, Xu Y, Zhang X, Bai C, Kang J, Ran P, Shen H, Wen F, Huang K, Yao W, Sun T, Shan G, Yang T, Lin Y, Wu S, Zhu J, Wang R, Shi Z, Zhao J, Ye X, Song Y, Wang Q, Zhou Y, Ding L, Yang T, Chen Y, Guo Y, Xiao F, Lu Y, Peng X, Zhang B, Xiao D, Chen CS, Wang Z, Zhang H, Bu X, Zhang X, An L, Zhang S, Cao Z, Zhan Q, Yang Y, Cao B, Dai H, Liang L, He J; China Pulmonary Health Study Group. Prevalence and risk factors of chronic obstructive pulmonary disease in China (the China Pulmonary Health [CPH] study): a national cross-sectional study. Lancet. 2018 Apr 28;391(10131):1706-1717. doi: 10.1016/S0140-6736(18)30841-9. Epub 2018 Apr 9. PMID 29650248
- See also: Global initiative for chronic obstructive lung disease.Global strategy for prevention,diagnosis and management of COPD — https://goldcopd.org/2024-gold-report/
- See also: Digital Therapeutics Alliance™.DTx Value Assessment & Integration Guide VERSION 2.0[EB/OL]（2022）[2024-7-26]. — https://dtxalliance.org/wp-content/uploads/2022/05/DTx-Value-Assessment-Guide_May-2022.pdf